CLINICAL TRIAL: NCT05861726
Title: Effects Of a Single Bout Of Acute Aerobic Exercise On Executive Brain Functions Of Young Adults: A Randomized Control Trial
Brief Title: Effects OF Acute Aerobic Exercise On Higher Cerebral Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khyber Medical College, Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 148/DME/KMC
Record Dates: First submitted 2023-03-14; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercising Group (Active Comparator): The exercising group shall have pre-intervention assessment of executive brain functions vide Stroop test, Trail making test & N-Back task/2-Back by using online psytoolkit followed by intervention.
  The intervention for the group being acute aerobic exercise, which will comprise of 30 minutes of treadmill walking at 60-65% of Heart Rate max with continuous recording of heart rate and ECG via Biopac MP36 Student Lab system.
  This will be followed by post-intervention assessment of executive brain functions vide Stroop test, Trail making test & N-Back task/2-Back by using online psytoolkit.
  Interventions: Behavioral: Aerobic exercise
- Control Group (Placebo Comparator): The control group will also have pre-intervention assessment of executive brain functions vide Stroop test, Trail making test & N-Back task/2-Back by using online psytoolkit.
  The control group will undergo NO EXERCISE intervention. They will sit idly in laboratory for 30 minutes with continuous recording of heart rate and ECG via Biopac system.
  The executive brain functions of the control group will be re-assessed vide Stroop test, Trail making test & N-Back task/2-Back by using online psytoolkit.
  Interventions: Other: None (control group)

INTERVENTIONS:
Behavioral: Aerobic exercise — a moderate kind of physical activity with a heart rate between 65 & 70% maximum heart rate
  Arms: Exercising Group
Other: None (control group) — None (the control group)
  Arms: Control Group

SUMMARY:
We are comparing higher cerebral functions including cognitive flexibility, inhibitory control and working memory in healthy young adults between a group of acute aerobic exercise and a control group.

DETAILED DESCRIPTION:
The objective of this study is to compare cognitive flexibility, inhibitory control, and working memory in healthy young adults between two groups: a group undergoing acute aerobic exercise and a control group.

Methodology:

Study Design: A Randomized Controlled Trial Study Setting: The Physiology Laboratory at Khyber Medical College, Peshawar Study Duration: The study will last for three months. Sample Size: The study will include 19 participants in each group - the Exercising group (E-Group) and the Control group (C-Group).

Healthy young people between 18-25 years who are non-smokers will be included. Sampling: The enrollment in the Randomised Control Trial will be conveniently based, wherein all those who meet the inclusion and exclusion criteria will be enrolled as per study numbers. A lottery method will be adopted for randomization.

Procedure:

The first step is to take ethical approval from the Institutional Research & Ethical Review Board. Following which, after taking informed consent from the participants, the enrolled participants will be randomly allocated to 2 groups. A demographic questionnaire will be filled. This will be followed by a general physical examination.

Both groups will be familiarized with the executive function tasks, while the E-group will have an additional session regarding the exercise protocol.

Both groups will have an initial assessment of executive functions using online psytoolkit followed by intervention. The E-group will undergo 30 minutes of treadmill walking at 60-65% of HRmax with continuous recording of heart rate and ECG via the Biopac system, while the control group session will consist of sitting idly and quietly in the laboratory doing nothing with continuous recording of heart rate and ECG via the Biopac student lab system.

In the end, executive function tests will be assessed before and after exercise using online psytoolkit.org. The data will be extracted via a properly designed proforma and on Microsoft Excel sheet.

Statistical Analysis:

Statistical Package for Social Sciences (SPSS)25.0 will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults

Exclusion Criteria:

* smokers
* cardiorespiratory disorders
* psychiatric disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in performance of Stroop Test before & after an acute session of aerobic exercise | Change in the reaction time of stroop test 5 minutes before and 3 minutes after aerobic exercise will be recorded
  Stroop test will be used to assess cognitive flexibility aspect of "executive brain functions".
  The reaction time in milliseconds to identify the congruent and incongruent words in the stroop test will be measured.
Change in performance of "Stop Signal Task Test" before & after an acute session of aerobic exercise. | Change in the response time 5 minutes before and 3 minutes after aerobic exercise will be recorded
  "Stop signal task" test will be used to assess the inhibitory control aspect of "executive brain functions".
  The response time in milliseconds will be measured in the test.
Change in performance of "Stop Signal Task Test" before & after an acute session of aerobic exercise. | Change in status of the response 5 minutes before and 3 minutes after aerobic exercise will be recorded
  "Stop signal task" test will be used to assess the inhibitory control aspect of "executive brain functions".
  Status of the response(1=correct, 2=wrong, 3=timeout) will be measured in the test.
Change in performance of "N-Back task/2-Back task " before & after an acute session of aerobic exercise. | Change in reaction time 5 minutes before and 3 minutes after an acute session of aerobic exercise will be recorded
  "N-Back task/2-Back task" test will be used to assess the working memory aspect of "executive brain functions".
  The reaction time taken in milliseconds to correctly match target letters in the test will be measured.
Change in performance of "N-Back task/2-Back task " before & after an acute session of aerobic exercise. | Change in the number of false alarms 5 minutes before and 3 minutes after an acute session of aerobic exercise will be recorded
  "N-Back task/2-Back task" test will be used to assess the working memory aspect of "executive brain functions".
  The number of false alarms on the test will be measured.

IPD SHARING:
Plan to Share IPD: No